CLINICAL TRIAL: NCT03794726
Title: A Prospective, Randomized Clinical Trial to Compare Orthodontic Molar Protraction With and Without Adjunctive Periodontally Accelerated Osteogenic Orthodontic (PAOO) Surgery.
Brief Title: Comparison of Orthodontic Molar Protraction With and Without Adjunctive Surgery
Acronym: PAOO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Maria L. Geisinger, DDS, MS, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-300002013; UAB-Perio (Other: University of Alabama at Birmingham)
Record Dates: First submitted 2018-10-09; First posted 2019-01-07 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Malocclusion
Keywords: Orthodontic tooth movement; Molar protraction; Periodontally accelerated osteogenic orthodontics; Patient-centered outcomes
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Orthodontic Molar Protraction (Active Comparator): Molar protraction using orthodontic tooth movement alone
  Interventions: Procedure: Orthodontic Molar Protraction
- Orthodontic Molar Protraction and PAOO (Experimental): Molar protraction using orthodontic tooth movement and adjunctive Periodontally Accelerated Osteogenic Orthodontics (PAOO)
  Interventions: Procedure: Orthodontic Molar Protraction and PAOO

INTERVENTIONS:
Procedure: Orthodontic Molar Protraction and PAOO — Molar Protraction with Orthodontic Tooth Movement and Adjunctive Periodontally Accelerated Osteogenic Orthodontics (PAOO) Surgery was performed on all study sites in this arm in coordination with standard orthodontic molar protraction using traditional bands/brackets and orthodontic wires.
  Arms: Orthodontic Molar Protraction and PAOO
Procedure: Orthodontic Molar Protraction — Standard orthodontic molar protraction using traditional bands/brackets and orthodontic wires.
  Arms: Orthodontic Molar Protraction

SUMMARY:
This study will compare orthodontic molar protraction with and without adjunctive periodontally accelerated osteogenic orthodontic (PAOO) surgery prior to orthodontic tooth movement.

To the investigators' knowledge, this type of molar retraction in adult patients has not been compared with and without the adjunctive use of PAOO for differences in clinical linear tooth movement and patient centered outcomes (discomfort, change in daily activities, satisfaction with esthetic outcomes) in a controlled study.

DETAILED DESCRIPTION:
Research data and daily clinical observations reveal that molar protraction (forward movement) in adult patients may be prolonged and ideal outcomes may not be achieved with traditional orthodontic tooth movement. One method for enhancing orthodontic tooth movement is the use of surgical access of the local site to initiate a regional tissue reaction to induce trauma, which leads to a limited inflammatory healing process. This process is also known as regional acceleratory phenomenon (RAP), which allows for more rapid bone turnover and has been shown in other protocols to enhance orthodontic tooth movement. While PAOO has been shown to rapidly increase tooth movement, to our knowledge, localized use of PAOO in combination with molar protraction in adults has not been evaluated in a prospective trial for differences in clinical outcomes (tooth movement time, adverse orthodontic outcomes, periodontal and soft tissue defects) and patient-centered outcomes (pain, swelling, change in daily activities, patient assessment of surgical benefit, and patient-assessed esthetics) in a controlled study.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* At least 18 years old
* Must be a patient of the University of Alabama at Birmingham (UAB) Dental School
* Able to read and understand informed consent document
* One or more nonadjacent 1st or 2nd molar teeth that require protraction of ≥ 5 mm in patients undergoing orthodontic tooth movement
* Presence of periodontally healthy, non-carious neighboring teeth, healthy implants or edentulous ridges on either side of the involved site(s)
* No anticipated need for restorative care at the teeth to be treated during the study period.

Exclusion Criteria:

* Non-English speaking
* Less than 18 years old
* Smokers/tobacco users (>10 cigarettes/day)
* Patients with systemic pathologies or conditions contraindicating oral surgical procedures or adversely affecting wound healing
* Presence of active periodontal disease, caries, and/or periapical pathology at teeth to be moved orthodontically
* Previous orthodontic therapy involving molar protraction of teeth to be treated
* Previous periodontal surgery at site(s) to be treated

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Linear millimeters of molar tooth movement | From baseline to 3months
  Compare the clinical linear molar tooth movement over a 3 month time frame (Baseline to 3 months) between two groups receiving orthodontic therapy alone or in combination with periodontally accelerated osteogenic orthodontics (PAOO).
Tooth angulation as measured radiographically | From baseline to 3months
  Compare the radiographic mesial inclination of the molar to be protracted over a 3-month time frame (Baseline to 3 months) between two groups receiving orthodontics therapy alone or in combination with periodontally accelerated osteogenic orthodontics (PAOO).

SECONDARY OUTCOMES:
Periodontal probing depth | From baseline to 3months
  Compare the periodontal probing depth (PD) at six sites per tooth at treated teeth over a 3-month time frame (Baseline to 3 months) between two groups receiving orthodontics therapy alone or in combination with periodontally accelerated osteogenic orthodontics (PAOO).
Periodontal clinical attachment level | From baseline to 3months
  Compare the clinical attachment level (CAL) at six sites per tooth at treated teeth over a 3-month time frame (Baseline to 3 months) between two groups receiving orthodontics therapy alone or in combination with periodontally accelerated osteogenic orthodontics (PAOO).
Periodontal width of keratinized tissue | From baseline to 3months
  Compare the width of keratinized tissue (KT) at up to two sites per tooth at treated teeth over a 3-month time frame (Baseline to 3 months) between two groups receiving orthodontics therapy alone or in combination with periodontally accelerated osteogenic orthodontics (PAOO).
Periodontal width of attached tissue | From baseline to 3months
  Compare the width of attached tissue at up to two sites per tooth at treated teeth over a 3-month time frame (Baseline to 3 months) between two groups receiving orthodontics therapy alone or in combination with periodontally accelerated osteogenic orthodontics (PAOO).
Practitioner-assessed treatment outcomes | From baseline to 3months
  Compare the practitioner-assessed esthetic outcomes using the pink esthetic score (PES) (Belser et al., 2009) over a 3-month time frame (Baseline to 3 months) between two groups receiving orthodontics therapy alone or in combination with periodontally accelerated osteogenic orthodontics (PAOO). This score is a grid which assesses mesial and distal papilla fill on a 0-2 scale, curvature of facial gingiva on a 0-2 scale, level of facial gingiva on a 0-2 scale, and root convexity/soft tissue color and contour on a 0-2 scale for an overall maximum assessment of 10 for esthetics. A 10 score would be considered ideal esthetics and a 0 would be considered least desirable. Each individual component of the PES is summed to provide the ultimate PES score.
Patient-assessed esthetic outcomes | From baseline to 3months
  Compare the patient-assessed satisfaction with esthetic outcomes over a 3-month time frame (Baseline to 3 months) between two groups receiving orthodontics therapy alone or in combination with periodontally accelerated osteogenic orthodontics (PAOO) using a visual analog scale from 0-100mm to determine the patients' assessment of their esthetic outcome.
Patient centered post-operative discomfort assessment | From baseline to 3months
  Compare treatment discomfort over a 3-month time frame (Baseline to 3 months) between two groups receiving orthodontics therapy alone or in combination with periodontally accelerated osteogenic orthodontics (PAOO) using a visual analog scale from 0-100mm to determine the patients' assessment of the post-operative discomfort.
Patient centered global treatment satisfaction | From baseline to 3months
  Compare treatment overall treatment satisfaction over a 3-month time frame (Baseline to 3 months) between two groups receiving orthodontics therapy alone or in combination with periodontally accelerated osteogenic orthodontics (PAOO) using a visual analog scale from 0-100mm to determine the patients' assessment of the patient's global assessment of treatment outcomes.
Patient centered alteration of daily activities assessment | From baseline to 3months
  Compare assessment of post-treatment change in daily activities over a 3-month time frame (Baseline to 3 months) between two groups receiving orthodontics therapy alone or in combination with periodontally accelerated osteogenic orthodontics (PAOO) using a visual analog scale from 0-100mm to determine the patients' assessment of the post-operative changes to daily activities.

CONTACTS AND LOCATIONS:
Overall Officials: Maria L Geisinger, DDS,MS, Principal Investigator — University of Alabama at Birmingham